CLINICAL TRIAL: NCT02018991
Title: Incidence and Predictors for Late Acquired Stent Malaposition of Drug-Eluting-Stents With Second-Generation Permanent and Biodegradable Polymer-Coatings - a Prospective, Randomized Comparison Using Optical Coherence Tomography
Brief Title: Late Acquired Malaposition and Different Polymers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Thomas Neunteufl, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUW-0001
Record Dates: First submitted 2013-12-17; First posted 2013-12-24 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Late Acquired Stent Malaposition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Everolimus-Eluting-Stent (EES) (Active Comparator): Patients treated with EES
  Interventions: Procedure: Everolimus-Eluting Stent (EES)
- Zotarolimus-Eluting-Stent (ZES) (Active Comparator): Patients treated with ZES
  Interventions: Procedure: Zotarolimus-Eluting-Stent (ZES)
- Biolimus-Eluting-Stent (BES) (Active Comparator): Patients treated with BES
  Interventions: Procedure: Biolimus-Eluting-Stent (BES)

INTERVENTIONS:
Procedure: Everolimus-Eluting Stent (EES) — Patients treated with EES
  Arms: Everolimus-Eluting-Stent (EES)
Procedure: Zotarolimus-Eluting-Stent (ZES) — Patients treated with ZES
  Arms: Zotarolimus-Eluting-Stent (ZES)
Procedure: Biolimus-Eluting-Stent (BES) — Patients treated with BES
  Arms: Biolimus-Eluting-Stent (BES)

SUMMARY:
The polymers releasing the drug of first-generation drug-eluting stents (DES) may induce allergic reactions and inflammation, resulting in late-acquired stent malaposition (LASM) with uncoverage of struts, and risk of stent thrombosis. The incidence and predictors of LASM in DES with newer-generation polymers designed to improve biocompatibility are unknown.

DETAILED DESCRIPTION:
please see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an elective treatment of a coronary lesion > 20mm with a DES

Exclusion Criteria:

* chronic renal failure (serum creatinine ≥ 2.5mg/dl)
* restenotic lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of stent struts with late acquired malaposition | 1 year after stent implantation

SECONDARY OUTCOMES:
number of stent struts with late acquired malaposition | 2 years after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neunteufl, Prof. Dr., Principal Investigator — PI
Locations (1):
- Medical University of Vienna, Vienna, Austria